CLINICAL TRIAL: NCT07270341
Title: Evaluation of Cerebral Oxygenation During Orthopedic Surgeries Performed in the Beach Chair Position Under General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nesil Coskunfirat, Prof Dr, Akdeniz University
Other Study IDs: TBAEK-727
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Perfusion; Cerebral Oxygenation; Hemodynamic Monitoring; Semi-sitting Position; Orthopedic Surgical Procedures
Keywords: cerebral perfusion; semi-sitting position; orthopedic surgery; cerebral oxygenation
MeSH Terms: interventions — Spectroscopy, Near-Infrared; Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic Surgery Patients in Semi-sitting Position: ASA I-III patients undergoing orthopedic surgery in the semi-sitting position, monitored with NIRS, invasive arterial pressure, and routine parameters.
  Interventions: Diagnostic Test: Near-Infrared Spectroscopy (NIRS) Monitoring

INTERVENTIONS:
Diagnostic Test: Near-Infrared Spectroscopy (NIRS) Monitoring — Cerebral oxygenation will be monitored using NIRS in addition to standard intraoperative monitoring (heart rate, invasive arterial pressure, end-tidal CO₂, and blood gas analysis).
  Other Names: Invasive Arterial Catheterization; Routine intraoperative monitoring including heart rate, non-invasive blood pressure, peripheral oxygen saturation, and end-tidal CO₂.

SUMMARY:
The goal of this observational study is to determine the correlation between cerebral oxygenation values measured by near-infrared spectroscopy (NIRS) and other routine monitoring parameters in patients placed in the semi-sitting position.

The primary questions investigated are :

Do NIRS values correlate with heart rate, invasive mean arterial pressure, and end-tidal carbon dioxide?

Do NIRS values reflect changes observed in arterial blood gas analysis?

Are cerebral perfusion-related parameters associated with patients' comorbidities such as diabetes, obesity, and hypertension?

Researchers will compare routine noninvasive monitoring (heart rate, blood pressure, peripheral oxygen saturation) with invasive arterial monitoring and NIRS to assess whether NIRS provides additional information for evaluating cerebral perfusion.

Participants will be monitored for:

Heart rate

Invasive mean arterial pressure

End-tidal carbon dioxide

Arterial blood gas changes

Cerebral oxygenation with NIRS

Patients' comorbidities (e.g., diabetes, obesity, hypertension) will also be recorded, and their association with perfusion-related parameters will be analyzed.

DETAILED DESCRIPTION:
Semi-sitting (beach chair) position is commonly used during orthopedic surgeries such as shoulder arthroscopy, clavicle fracture fixation, and proximal humerus operations. However, this position is associated with a risk of cerebral hypoperfusion due to gravitational redistribution of blood volume, leading to decreased mean arterial pressure at the brain level. This can result in severe complications such as visual loss, ischemic stroke, and even brain death.

Routine noninvasive monitoring methods, including heart rate, blood pressure, and peripheral oxygen saturation, are standard during anesthesia. Because of the frequent occurrence of hypotension in this position, invasive arterial pressure monitoring is recommended to detect and manage hemodynamic fluctuations more precisely. Near-infrared spectroscopy (NIRS) is a noninvasive method that allows continuous measurement of cerebral oxygenation and can identify early reductions in cerebral perfusion that may not yet be reflected in traditional monitoring parameters.

The aim of this prospective observational cohort study is to determine the correlation between cerebral oxygenation measured by NIRS and other hemodynamic parameters (heart rate, invasive mean arterial pressure, end-tidal carbon dioxide) as well as arterial blood gas analysis during orthopedic surgery performed in the semi-sitting position. Additionally, the study will evaluate the relationship between cerebral perfusion parameters and patients' comorbidities (e.g., diabetes, hypertension, obesity, and other chronic conditions) to identify potential risk factors for cerebral desaturation in this surgical position.

The study will be conducted in a single tertiary academic center. A total of 30 adult patients (ASA I-III), aged 18 years or older, scheduled for elective orthopedic surgery in the semi-sitting position will be enrolled. Standard anesthesia care will be applied to all patients, and no additional intervention will be performed beyond routine monitoring. Data collection will include continuous NIRS measurements, invasive arterial pressure, heart rate, peripheral oxygen saturation, end-tidal CO₂, and arterial blood gas results.

Statistical analysis:

Descriptive statistics will be presented as means and standard deviations for continuous variables, and frequencies for categorical variables. Normality will be assessed using the Kolmogorov-Smirnov test. Correlations between NIRS values and other parameters (mean arterial pressure, ETCO₂, heart rate, blood gas values) will be analyzed using Pearson correlation coefficients for normally distributed variables. Group comparisons will be performed using paired t-tests for parametric data and Mann-Whitney U tests for nonparametric data. Bonferroni correction will be applied where multiple comparisons are made. A p-value of <0.05 will be considered statistically significant.

Sample size was calculated using G*Power (version 3.1.9.7) with a power of 80%, alpha of 0.05, and a medium effect size (f=0.25), resulting in a minimum of 28 patients required. Data will be analyzed using SPSS version 15.0.

This study aims to contribute to identifying optimal intraoperative monitoring strategies for maintaining cerebral perfusion during orthopedic procedures performed in the semi-sitting position, particularly in patients with multiple comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for orthopedic surgery in the semi-sitting position
* ASA physical status I-III
* Voluntary participation with informed consent

Exclusion Criteria:

* Patients younger than 18 years
* Patients who do not provide consent
* History of cerebral ischemia
* History of head trauma
* Previous neurosurgical intervention
* Documented carotid stenosis ≥90%
* Previous neck surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years and older, ASA I-III) undergoing orthopedic surgery in the semi-sitting position, monitored for cerebral oxygenation (NIRS), invasive arterial pressure, and routine intraoperative parameters.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Cerebral Oxygenation (rSO₂) Measured by NIRS and Systemic Oxygenation | From pre-induction baseline through post-induction and positional measurements, followed by repeated assessments every 30 minutes until the end of surgery.
  The correlation between intraoperative cerebral oxygenation (regional cerebral oxygen saturation, rSO₂) (%)-measured non-invasively using near-infrared spectroscopy (NIRS) -and simultaneous systemic oxygenation assessed using arterial blood gas analysis, including: Arterial pH, PaO₂ (mmHg) and PaCO₂ (mmHg)
Correlation Between Cerebral Oxygenation (rSO₂) Measured by NIRS and Hemodynamic Parameters (Heart Rate and Blood Pressure) | From pre-induction baseline through post-induction and positional measurements, followed by repeated assessments every 30 minutes until the end of surgery.
  The correlation between intraoperative cerebral oxygenation (regional cerebral oxygen saturation, rSO₂) (%)-measured non-invasively using near-infrared spectroscopy (NIRS) -and systemic hemodynamic parameters.
  Systemic hemodynamic parameters will include:
  1. Heart rate (beats per minute), monitored continuously via electrocardiography (ECG)
  2. Noninvasive mean arterial pressure (mmHg), measured using an automated oscillometric device
  3. Invasive mean arterial pressure (mmHg), obtained via an arterial catheter

SECONDARY OUTCOMES:
Association of Preoperatively Documented Hypertension with Intraoperative Low Cerebral Oxygenation (rSO₂) Measured by Near-Infrared Spectroscopy | Preoperative period for comorbidity assessment and intraoperative period for cerebral oxygenation measurements (from pre-induction baseline to the end of surgery.
  The associations between preoperatively diagnosed hypertension with the occurrence of intraoperative reductions in regional cerebral oxygen saturation (rSO₂), defined as values falling below the normal range (60-75%).
Association of Preoperatively Documented Diabetes Mellitus with Intraoperative Low Cerebral Oxygenation (rSO₂) Measured by Near-Infrared Spectroscopy | Preoperative period for comorbidity assessment and intraoperative period for cerebral oxygenation measurements (from pre-induction baseline to the end of surgery.
  The associations between preoperatively diagnosed diabetes mellitus, and the occurrence of intraoperative reductions in regional cerebral oxygen saturation (rSO₂), defined as values falling below the normal range (60-75%).
Association of Preoperatively Documented Obesity with Intraoperative Low Cerebral Oxygenation (rSO₂) Measured by Near-Infrared Spectroscopy | Preoperative period for comorbidity assessment and intraoperative period for cerebral oxygenation measurements (from pre-induction baseline to the end of surgery.
  The associations between preoperative obesity-defined as a body mass index (BMI) greater than 30 kg/m²-and the occurrence of intraoperative reductions in regional cerebral oxygen saturation (rSO₂), defined as values falling below the normal range (60-75%).

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu S, Bloomquist D. Can resorbable screws effectively be used in fixating bilateral sagittal split osteotomies for mandibular advancement? A randomized controlled trial. J Oral Maxillofac Surg. 2014 Nov;72(11):2273-7. doi: 10.1016/j.joms.2014.04.033. Epub 2014 May 9. PMID 25086478
- [Background] Carroll JJ, Marshall BDL, Rich JD, Green TC. Exposure to fentanyl-contaminated heroin and overdose risk among illicit opioid users in Rhode Island: A mixed methods study. Int J Drug Policy. 2017 Aug;46:136-145. doi: 10.1016/j.drugpo.2017.05.023. Epub 2017 Jun 1. PMID 28578864